CLINICAL TRIAL: NCT05279469
Title: D-Dimer as Predictor of Disease Outcome in Intensive Care Unit in SARS-COV-2 Patients: A Retrospective Study
Brief Title: D-Dimer as Predictor of Disease Outcome in Intensive Care Unit in COVID-19m Patients
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amr M Hilal Abdou, Assistant Professor, Ain Shams University
Other Study IDs: MS56/2022
Record Dates: First submitted 2022-03-10; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Critical Illness; Pneumonia, Viral
Keywords: D dimer; SARS-COV-2
MeSH Terms: conditions — Critical Illness; Pneumonia, Viral | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention, just observational for D-Dimer level in blood — observation for basal D-Dimer and 48 hours later D-Dimer in blood for ICU SARS.COV.2 patients

SUMMARY:
Evaluating value of D-Dimer blood level of icu admitted patients on admission and 48 hours later as outcome predictor in SARS.COV.2 patients.

DETAILED DESCRIPTION:
Evaluating value of D-Dimer blood level of icu admitted patients on admission and 48 hours later as outcome predictor in SARS.COV.2 patients.

It has been reported that COVID 19 is associated with hemostatic abnormalities and elevated D-Dimer level, so its level is used to predict severity of disease.

ELIGIBILITY:
Inclusion Criteria:

* patients of both sex admitted in icu
* positive PCR
* requiring oxygen therapy

Exclusion Criteria:

* ward patients
* negative PCR

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients in SARS.COV.2 patients in ICU with positive PCR and needing oxygen therapy
Sampling Method: Non-Probability Sample
Enrollment: 465 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
28 days mortality | 1 month
  Outcomes of ICU stay

SECONDARY OUTCOMES:
length of stay and mechanical ventilation | during ICU stay
  time of admission and need to escalate oxygen therapy

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ain shams university hospitals, Cairo
  - Faculty of medicine, Ain Shams University, Cairo

IPD SHARING:
Plan to Share IPD: Undecided